CLINICAL TRIAL: NCT05841602
Title: Quality of Nursing Care During The Covid-19 Pandemic From The Perspective Of Hospitalized Children: A Cross-Sectional Study
Brief Title: Quality of Nursing Care During The Covid-19 Pandemic
Status: Completed | Type: Observational
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Mukaddes Demir Acar, Ass. Prof., Tokat Gaziosmanpasa University
Other Study IDs: MDEMIRACAR
Record Dates: First submitted 2023-04-29; First posted 2023-05-03 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-05

CONDITIONS: COVID-19 Pandemic; Children, Only; Hospitalism; Nurse's Role; Feelings
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- study group: 8-13 age group (N=128).
  Interventions: Other: descriptive

INTERVENTIONS:
Other: descriptive — This research was conducted to evaluate nursing care from the perspective of hospitalized children during the Covid-19 pandemic process and to determine their feelings during this process.

SUMMARY:
Enabling school-age children to evaluate the care they receive provides feedback on the quality of care by determining children's satisfaction with care, and gives important feedback on the quantity and quality of care. Evaluation of nursing care, emotions and behaviors from the perspective of children during the Covid-19 pandemic process will guide the improvement of the quality of care. As a result of the literature review on this subject, no research has been found, and it is thought that this research will contribute to the field. This research was conducted to evaluate nursing care and emotions from the perspective of hospitalized children during the Covid-19 pandemic process.

ELIGIBILITY:
Inclusion Criteria:

* The study included volunteer children who were hospitalized for at least 3 days in the - -- -pediatric clinic,
* whose native language was Turkish,
* between the ages of 8-13,
* who did not have any visual, auditory or mental problems, and whose parents gave consent for the study.

Exclusion Criteria:

* who fall outside the inclusion criteria

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: This cross-sectional descriptive study was conducted in a hospital in the Black Sea Region of XXX between February and June 2021
Sampling Method: Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
The Scale Evaluation Quality of Care From Children's Point of View | 4 month
  The Scale Evaluation Quality of Care From Children's Point of View is a 5-point Likert-type scale (never = 1, rarely agree = 2, sometimes agree= 3, often agree = 4, always agree=5) involving 15 items, which was developed by Yilmaz and Ak (2018). The minimum score that can be obtained from the scale is 15 and the maximum score is 75.

CONTACTS AND LOCATIONS:
Overall Officials: Mukaddes Demir Acar, Study Chair — Tokat Gaziosmanpasa University
Locations (1):
- Tokat Gaziosmanpasa University, Tokat Province, Eyalet/Yerleşke, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: SAP